CLINICAL TRIAL: NCT03451643
Title: Comparison Between Endoscopic Stenting and Colorectal Resection in Patients With Stage IV Colorectal Cancer
Brief Title: Stenting and Resection for Stage IV Colorectal Cancer Endoscopic Stenting and Colorectal Resection in Stage IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, antonio sterpetti, AGGREGATE PROFESSOR OF SURGERY, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1010236
Record Dates: First submitted 2017-04-27; First posted 2018-03-02 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Neoplasm
Keywords: colorectal cancer; liver metastases; stage IV
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: RANDOMIZED CONTROLLED TRIAL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Expandable Stent (Experimental): Procedure/Surgery. Endeosocpically a self-expandable metal stent will be placed in the colon rectum. Chemotherapy will be added
  Interventions: Procedure: ENDOSCOPIC PLACEMENT OF EXPANDABLE STENT
- Colorectal Resection (Active Comparator): Procedure/Surgery. A standard open or laparoscopic surgery will be performed to remove the colorectal cancer. Chemotherapy will be added
  Interventions: Procedure: ENDOSCOPIC PLACEMENT OF EXPANDABLE STENT

INTERVENTIONS:
Procedure: ENDOSCOPIC PLACEMENT OF EXPANDABLE STENT — PLACEMENT OF AN ENDOSCOPIC SELF EXPANDABLE METAL STENT
  Other Names: CHEMOTHERAPY

SUMMARY:
Patients with Stage IV obstructing colorectal cancer and unresectable liver metastses, with general and local conditions not a risk for coliorectal resection, will be randomized to have either endoscopic stenting or colorectal resection

DETAILED DESCRIPTION:
Patients with obstructing colorectal cancer, Stage IV with not resectable metastases will be considered .

Patients with acceptable general and local conditions, to allow a safe surgical resection will be considered.

Patients will be randomized to have endoscopic stenting or colorectal resection.

All patients will receive postoperative chemio therapy

ELIGIBILITY:
Inclusion criteria

* Patients with Stage IV obstructing colorectal cancer and liver metastases
* Liver metastases not resectable

Exclusion criteria

-Patients considered at high risk for colorectal resection

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
MORTALITY | 60 DAYS
  THE NUMBER OF POSTPROCEDURAL DEATHS
SURVIVAL | 5 YEARS
  SURVIVAL IN MONGTHS WILL BE DETERMINED FOR PATIENTS USING KAPLAN MEIER CURVES AND MEDIAN SURVIVAL
POSTOPERATIVE MORBIDITY | 60 DAYS
  MAJOR AND MINOR COMPLICATIONS AFTER THE PROCEDURE

SECONDARY OUTCOMES:
QUALITY OF LIFE | 5 YEARS
  QUALITY OF LIFE WILL BE ASSESSED USING A STANDARDIZED PROTOCOL

CONTACTS AND LOCATIONS:
Overall Officials: antonietta lamazza, MD, Study Director — University of Rome
Locations (2):
- Italy (2):
  - Istituto Pietro Valdoni, Rome
  - University of Rome Sapienza, Rome

IPD SHARING:
Plan to Share IPD: Yes
IPD data will be shared with publications and conferebnces
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 10.02.2018 for 3 months
Access Criteria: contact by e-mail